CLINICAL TRIAL: NCT01349985
Title: SBIR-PhaseII, "Adaptive Goal-Directed Adherence Tracking and Enhancement"
Brief Title: Adaptive Goal-Directed Adherence Tracking and Enhancement
Acronym: AGATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Talaria, Inc (Industry)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HHSN275201000011C; HHSN275201000011C (Other: NIAAA SBIR Contract)
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Alcohol Abuse
Keywords: Naltrexone; problem drinking; medication adherence; adherence; smartphone
MeSH Terms: conditions — Alcoholism; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AGATE (Experimental): To evaluate whether AGATE, a smartphone medication reminder and assessment system, effectively measures and enhances medication adherence in the context of naltrexone treatment for problem drinking.
  Interventions: Other: AGATE
- SASED (Active Comparator): The control condition for the proposed study is a smartphone alcohol and side-effects diary (SASED, a smartphone alcohol and side effects diary).
  Interventions: Other: SASED

INTERVENTIONS:
Other: AGATE — AGATE is a web-based adherence-enhancement intervention accessible via smartphone. All participants will be prescribed naltrexone, 50 mg, once daily for eight weeks.
  Arms: AGATE
Other: SASED — Participants will receive SASED, a web-based alcohol and side-effects diary via smartphone. All participants will be prescribed naltrexone, 50 mg, once daily for eight weeks.
  Arms: SASED

SUMMARY:
Talaria, Inc., has designed an adherence tracking and enhancement system, called AGATE, which uses the text messaging and internet capabilities of modern cellular phones to address the problem of medication adherence in clinical care and clinical trial contexts. This trial will evaluate whether AGATE improves medication adherence in the context of a pharmacotherapy trial of naltrexone to treat problem drinking. All participants will be treatment-seeking problem drinkers who will receive naltrexone and medication monitoring over 8 weeks.

DETAILED DESCRIPTION:
The purpose of the naltrexone trial is to evaluate whether AGATE effectively measures and enhances medication adherence in the context of naltrexone treatment for problem drinking. Participants will be heavy/problem drinkers, recruited from the greater Albuquerque area, who are interested in either reducing or stopping their drinking and deemed to be candidates for naltrexone pharmacotherapy by the study psychiatrist, Dr. Arenella. All participants will be prescribed naltrexone, 50 mg, once daily, for eight weeks, and receive smartphones. Participants will be randomly assigned to receive either AGATE or SASED, a web-based alcohol and side-effects diary via smartphone. The primary outcome will be percent of scheduled doses that were taken during the eight week trial, as measured by the Medication Event Monitoring System (MEMS, Aardex Group, Union City, CA), pill counts, and using the timeline follow-back (TLFB) method.

ELIGIBILITY:
Inclusion Criteria:

* problem or heavy drinkers
* age 21-55 years old
* located in the greater Albuquerque NM area
* interested in either reducing or stopping their drinking
* candidates for naltrexone pharmacotherapy

Exclusion Criteria:

* participation in other naltrexone study
* unable to operate a smartphone
* significant psychiatric or physical illness
* current drug dependence
* current regular opioid use
* any recent nonmedical opioid use
* any lifetime opioid dependence

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2011-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 8 weeks
  Adherence will be measured using the medication event monitoring system (MEMS), pill counts, and multiple self-report indices.

SECONDARY OUTCOMES:
Indices of alcohol use, craving, etc. | 8 weeks
  Indicies of alcohol use, cravings etc will be measured using validated patient self report measures.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Stoner, Ph.D., Principal Investigator — Talaria, Inc
Locations (1):
- The Mind Research Network, University of New Mexico, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Stoner SA, Arenella PB, Hendershot CS. Randomized controlled trial of a mobile phone intervention for improving adherence to naltrexone for alcohol use disorders. PLoS One. 2015 Apr 24;10(4):e0124613. doi: 10.1371/journal.pone.0124613. eCollection 2015. PMID 25909320
- [Derived] Stoner SA, Hendershot CS. A randomized trial evaluating an mHealth system to monitor and enhance adherence to pharmacotherapy for alcohol use disorders. Addict Sci Clin Pract. 2012 Jun 8;7(1):9. doi: 10.1186/1940-0640-7-9. PMID 23186301